CLINICAL TRIAL: NCT01085292
Title: NOX-E36 - A Phase Ib, Multiple Intravenous Dose Study to Evaluate Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Properties in Healthy Subjects and Then in Three Groups of Patients With Type 2 Diabetes Mellitus to Compare Three Ascending Dose Regimens in a Double-blind and Placebo-controlled Manner
Brief Title: NOX-E36 Multiple Ascending Dose Study in Healthy Volunteers and Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TME Pharma AG (Industry)
Collaborators: Profil Institut für Stoffwechselforschung GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: SNOXE36C101; 2010-019148-38 (EudraCT Number)
Record Dates: First submitted 2010-03-10; First posted 2010-03-11 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental)
  Interventions: Drug: NOX-E36
- Group B - D (Experimental)
  Interventions: Drug: NOX-E36

INTERVENTIONS:
Drug: NOX-E36 — Multiple dose 0.25 mg/kg or placebo i.v. to healthy volunteers; dosing frequency q2d
  Arms: Group A
Drug: NOX-E36 — Multiple dose of 0.0625 mg/kg, 0.125 mg/kg, 0.25 mg/kg or placebo i.v. to patients with type 2 diabetes mellitus (ratio 3:1); dosing frequency q2d
  Arms: Group B - D

SUMMARY:
The primary objective of this trial is to evaluate the safety and tolerability of multiple intravenous doses of NOX-E36 in healthy subjects and patients with type 2 diabetes mellitus. A secondary objective of the trial is to obtain exploratory estimates of the pharmacodynamic response at the level of inflammation, metabolism as well as ongoing diabetes complications (e.g. impaired cardiovascular, liver and renal function). Thus, the study is designed to provide sufficient safety and dose-response data for a planned Phase IIa proof of concept study with NOX-E36 in patients with multiple complications of type II diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Group A: Healthy male and female subjects
* Group B-D: Patients with type 2 diabetes mellitus according to ADA definition; GFR > 60 mL/min; HbA1c ≥ 6.0 and ≤9.0 %; normoalbuminuria, microalbuminuria or macroalbuminuria

Exclusion Criteria:

* History of or presence of clinically significant diseases with the exception of diabetes (Groups B-D)
* Concurrent illness that may affect blood glucose other than diabetes
* Supine blood pressure at screening, after resting for 5 min, of >140 mmHg systolic or > 90 mmHg diastolic (Group A) or > 160 mmHg systolic or > 95 mmHg in diabetes mellitus patients (Groups B-D)
* Clinically significant abnormal ECG at screening
* Any kidney disease not caused by diabetes or hypertension
* Type 1 diabetes mellitus

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2010-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of multiple intravenous doses of NOX-E36 in healthy subjects and patients with type II diabetes mellitus | 4 weeks

SECONDARY OUTCOMES:
Multiple dose pharmacokinetics and pharmacodynamics of NOX-E36 in healthy subjects and patients with type II diabetes mellitus | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Grit Landgraf, PhD, Study Director — Noxxon AG
Locations (5):
- Germany (5):
  - Itecra GmbH, Cologne
  - CTC North MediGate GmbH, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - ikfe GmbH, Mainz
  - Profil Institut fuer Stoffwechselforschung GmbH, Neuss

REFERENCES:
- [Derived] Park EJ, Choi J, Lee KC, Na DH. Emerging PEGylated non-biologic drugs. Expert Opin Emerg Drugs. 2019 Jun;24(2):107-119. doi: 10.1080/14728214.2019.1604684. Epub 2019 Apr 19. PMID 30957581